CLINICAL TRIAL: NCT06080607
Title: Rehabilitation Needs in Patients With Early Breast Cancer: Validation of a Questionnaire Patient Reported Outcome
Brief Title: PRO Survivorship Concerns ITA
Acronym: PRO
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Centro di Riferimento Oncologico - Aviano (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); Istituti Tumori Giovanni Paolo II (Network); Fondazione Salvatore Maugeri (Other)
Responsible Party: Sponsor
Other Study IDs: RS1272/19
Record Dates: First submitted 2023-03-24; First posted 2023-10-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Breast Neoplasm Female; Quality of Life; Psychological Distress
MeSH Terms: interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Patient Reported Outcome (PRO) — Quality of Life evaluation

SUMMARY:
Breast cancer survivors typically experience fatigue, pain, insomnia, depression, anxiety, difficulty in concentrating, memory impairment, body image problems, vaginal dryness, interest in sex decreasing, hot flashes, gain weight, and infertility. All of these problems affect quality of life (QoL) mainly during the early survival and they become even more important to understand and address if long-term effects could be prevented.

The use of PROs in care settings has demonstrated improvement in provider/patient communication, recognition of previously unrecognized issues, as well as patient satisfaction with care.

In order to allow to patients the use of the PRO "survivorship concerns" in their mother tongue, it is imprtant to have validated translations with transcultural adaptation. The main goals of this multicentric study are the translation, adaptability and transcultural validation of the PRO questionnaire "survivorship concerns" to put in evidence rehabilitation needs in breast cancer patients in early stage.

ELIGIBILITY:
Inclusion Criteria:

* During transcultural adaptability 80 representative patients will be recruited .

During the validation phase previus patients will be included and more other patients will be included (at least 280)

Exclusion Criteria:

* Patients with cognitive or memory impairment wil be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer women patients
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-06-18 (Estimated); Study Completion 2024-06-18 (Estimated)

PRIMARY OUTCOMES:
Translation and validation of questionnaire PRO | 6 months
  The main goals of this multicentric study are the translation, adaptability and transcultural validation of the PRO questionnaire "survivorship concerns" to put in evidence rehabilitation needs in breast cancer patients in early stage.
  the PRO questionnaire "survivorship concerns" is made up of 17 items which evaluate the problems of survival, the level of concern about problems related to the care of patients, screening, symptom management, family and genetic problems and the fear of disease recurrence, on a scale of 0 to 3.It will be administered twice 15 days apart and in order to identify the levels of agreement between the two assessments, the Interclass Correlation Coefficient (ICC) model 3.1 will be applied and calculated for each item.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Regina Elena Cancer Institute, Rome, Roma
  - "Regina Elena" National Cancer Institute, Rome

IPD SHARING:
Plan to Share IPD: Undecided